CLINICAL TRIAL: NCT01426139
Title: BIOTRONIK-Safety and Clinical PerFormance of the Drug Eluting ORSIRO Stent in the Treatment of Patients With Single de Novo Coronary Artery Lesions in an Indian Population
Brief Title: BIOFLOW-INDIA Safety and Clinical PerFormance of the Drug Eluting ORSIRO Stent in Single de Novo Coronary Artery Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C1002
Record Dates: First submitted 2011-08-10; First posted 2011-08-31 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biotronik Orsiro DES (Experimental)
  Interventions: Device: Percutaneous Coronary Intervention Biotronik Orsiro DES

INTERVENTIONS:
Device: Percutaneous Coronary Intervention Biotronik Orsiro DES — Stenting

SUMMARY:
The objective of this clinical investigation is to assess the safety and clinical performance of the Orsiro Limus Eluting Stent System in Indian subjects with single de-novo coronary artery lesions.

ELIGIBILITY:
Main Inclusion Criteria:

* Subject has provided a written informed consent
* Single de novo lesion with ≥ 50% and <100% stenosis in up to 2 coronary arteries
* The target lesion length is ≤ 26 mm
* The target reference vessel diameter is ≥ 2.0 mm and ≤ 4.0 mm

Main Exclusion Criteria:

* Evidence of myocardial infarction within 72 hours prior to index procedure
* Unprotected left main coronary artery disease (stenosis >50%)
* Three-vessel coronary artery disease at time of procedure Thrombus in target vessel
* Target lesion involves a side branch > 2.0 mm in diameter
* Heavily calcified lesion
* Target lesion is located in or supplied by an arterial or venous bypass graft

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2011-08; Primary Completion 2012-11 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
In-Stent Late Lumen Loss | 9 months post index procedure

CONTACTS AND LOCATIONS:
Locations (4):
- India (4):
  - Madras Medical Mission, Chennai
  - Medanta The Medicity Hospital, Gūrgaon
  - Max Super Speciality Hospital, New Delhi
  - Fortis Escorts Heart Institute and Research Centre, New Delhi